CLINICAL TRIAL: NCT06532734
Title: Presence of Barrett's Esophagitis in a Cohort of People With Eating Disorders Who Engage in Purging Behaviors: A Pilot Study
Brief Title: Barrett's Esophagitis in Anorexia Nervosa Binge/Purge Subtype
Status: Recruiting | Type: Observational
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Lucid Diagnostics, Inc. (Industry)
Responsible Party: Principal Investigator, Allison Nitsch, Lead Hospitalist, Denver Health and Hospital Authority
Other Study IDs: 24-0349
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Barrett Esophagus; Anorexia Nervosa, Binge Eating/Purging Type; Rumination; Vomiting; Eating Disorders; Esophageal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Anorexia Nervosa; Bulimia; Rumination Syndrome; Vomiting; Feeding and Eating Disorders; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- AN-BP: individuals with a dx of AN-BP, with a >5-year history of purging, with a frequency of at least once a day.
  Interventions: Device: EsoGuard

INTERVENTIONS:
Device: EsoGuard — device used to collect esophageal cell samples to test for the presence of abnormal cells which may indicate a dx of Barrett's esophagitis.

SUMMARY:
To better define the presence of Barrett's esophagus (BE) via non-endoscopic testing in an eating disorder cohort with purging (vomiting/rumination) behaviors

DETAILED DESCRIPTION:
A prospective cohort study to assess the presence of BE in those with purging behaviors from their eating disorders has not been completed. There are multiple case reports describing a younger population not meeting typical screening guidelines whom developed this condition. To better define the presence of Barrett's esophagus (BE) via non-endoscopic testing in an eating disorder cohort with purging (vomiting/rumination) behaviors. Individuals with severe forms of eating disorders with purging and ruminating behaviors not meeting the current screening guidelines for BE will still test positive for BE.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with an eating disorder diagnosis that includes purging history
* Ages 18-65
* Purging history =>5 years
* Purging or rumination at a minimum of once daily upon admission.
* Admission to the ACUTE Center for Eating Disorders and Severe Malnutrition

Exclusion Criteria:

* Any eating disorder diagnosis that does not include purging behaviors
* Ages under 18 and over 65
* Patients who otherwise meet the current ACG screening guidelines (chronic GERD and 3 or more risk factors for Barrett's mentioned in the Background)
* Received mandated care at time of enrollment
* Inability to consent to participate in the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACUTE patients with a confirmed dx of AN-BP, with a purging history of >5 year, with a frequency of purging of at least once a day.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients positive for BE | 12 months
  Individuals with severe forms of eating disorders with purging and ruminating behaviors not meeting a current screening guidelines for BE will test positive for BE

CONTACTS AND LOCATIONS:
Overall Officials: Allison Nitsch, MD, Principal Investigator — Denver Health and Hospital Authority
Locations (2):
- United States (2):
  - ACUTE Center for Eating Disorders and Severe Malnutrition, Denver, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No